CLINICAL TRIAL: NCT02002780
Title: Recognizing and Treating Psychosocial Stress Among Children With Complex Heart Problems
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study not started, investigator left the institution
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Brian McCrindle, Staff Cardiologist, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000020209
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-12

CONDITIONS: Psychosocial Stress
Keywords: pediatrics; stress; cardiac surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subjects (Experimental): Children identified during the screening phase of the project as having elevated, but not clinically defined, levels of psychosocial stress will be invited to participate in the intervention phase of this research if they are between 8 and 11 years of age.
  Screening will identify 6 girls and 6 boys eligible and willing to participate in the intervention phase of the project.
  Interventions: Behavioral: Day Camp
- Control (No Intervention): All families that were screened during the screening phase of this study will complete the final screening instrument assessment, whether or not the child participated in the day camp intervention. The control group will be comprised of those families that did not participate in the intervention.

INTERVENTIONS:
Behavioral: Day Camp — The intervention will be delivered using a day camp structure, on a weekend or during school break in July 2011. Separate interventions will be offered for boys and girls. Each intervention will include two full days (0900 to 1600) of group activities lead by the researchers. Details of the "camp" activities will be developed by the researchers, based on the types of psychosocial stress identified during the screening phase of the project.
  Arms: Subjects

SUMMARY:
This research project has two goals. The first goal is to find one or more questionnaires that can accurately identify children who are experiencing high levels of stress or emotional health issues during a regular clinic visit. The second goal is to find out whether children who are experiencing stress or emotional health problems are able to attend a day camp programme and complete activities at home that are designed to help them cope better with stress. We also want to find out if the day camp and home activities are helpful.

DETAILED DESCRIPTION:
This research will investigate the psychological stress experienced by children who have had surgery for a complex heart problem. Measures of quality of life among children with heart problems indicate that those 8 to 12 years of age have lower quality of life scores than younger or older children.

Children who survive a critical illness requiring a multi-day stay in a pediatric intensive care unit are at risk for a variety of psychiatric morbidities. Depression, anxiety and post-traumatic stress disorder occur in 7% to 28% of patients.

A systematic review of psychological adjustment among children with heart problems indicates that parent reports (but not child self-reports) are useful in detecting problems with psychological adjustment. While parent reports tend to identify increased social and behaviour problems, child self-reports indicate more frequent symptoms of depression compared to healthy peers.

ELIGIBILITY:
Inclusion Criteria:

* children who have had surgery for a complex heart problem
* children with heart problems requiring on-going medical care
* age 6 to 12 years

Exclusion Criteria:

* the child has had an intervention (catheterization or surgery) within the previous 6 months,
* the child has an identified cognitive or emotional health disability,
* the child or parents do not speak English sufficiently well to respond to the screening instruments, or
* the child's clinic visit is for an acute illness or change in health status.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Change in psychosocial stress scores resulting from the intervention | Baseline and end of study (at about month 10 -11)

CONTACTS AND LOCATIONS:
Overall Officials: Brian McCrindle, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada